CLINICAL TRIAL: NCT06464640
Title: Efficacy of the Interactive Podcast Program "Living With Type 1 Diabetes to Grown-Up": A Two-arm Randomized Controlled Trial
Brief Title: Efficacy of the "Living With Type 1 Diabetes to Grown-Up" Interactive Podcast Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yueh-Tao Chiang, Assistant Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: T1dPodcastchanggungU
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; transition; podcast; self-regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Self-Control

STUDY DESIGN:
Intervention Model Description: Experimental group: The Online Interactive Podcast Program"Living with Type 1 Diabetes to Grown-Up" will be used for intervention in the experimental group.
  active control group:E-book.According to the research results from the project Healthcare CEO app effectiveness evaluation (Chiang, 2020-2022), the e-book did not show significant effects on blood sugar control, disease management confidence, self-care behaviors, disease-related knowledge, or interpersonal distress. Therefore, the active control group received a sham treatment in the form of an e-book. The research team extracted content from the CEO APP e-book, with an expert validity of 0.91, and reorganized it into an electronic health education manual titled"Transitioning from Adolescence to Early Adulthood: The Ins and Outs of Type 1 Diabetes."
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- podcast intervention (Experimental): The podcast will be used for intervention in the experimental group.
  Interventions: Device: Online Interactive Podcast Program "Living with Type 1 Diabetes to Grown-Up"
- Ebook intervention (Sham Comparator): Participants in the active control group will use E-book.
  Interventions: Device: E-book

INTERVENTIONS:
Device: Online Interactive Podcast Program "Living with Type 1 Diabetes to Grown-Up" — The podcast content was designed based on the results of previous research.Subjects will be randomly assigned to either the experimental group (N=44) or the comparison group (N=44). Comparative analyses will focus on variations in disease control, emotional disturbance,confidence in self-management, self-care behaviors, diabetes knowledge,interpersonal disturbance, and family conflict at baseline, and post-interventions of immediate, 3-month, and 6-month periods.
  Arms: podcast intervention
Device: E-book — Participants in the active control group will use Ebook.According to the research results from the project leader's app effectiveness evaluation (Chiang, 2020-2022), the e-book did not show significant effects on blood sugar control, disease management confidence, self-care behaviors, disease-related knowledge, or interpersonal distress. Therefore, the active control group received a sham treatment in the form of an e-book. The research team extracted content from the CEO APP e-book, with an expert validity of 0.91, and reorganized it into an electronic health education manual titled "Transitioning from Adolescence to Early Adulthood: The Ins and Outs of Type 1 Diabetes."
  Arms: Ebook intervention

SUMMARY:
The present study aims to evaluate the intervention effectiveness of the Online Interactive Podcast Program"Living with Type 1 Diabetes to Grown-Up"in patients with type 1 diabetes transitioning from adolescence to early adulthood.

DETAILED DESCRIPTION:
Individuals aged 16-25 with Type 1 Diabetes (T1D) face significant transitional challenges in their lives, with an increased risk of worsening disease management. Addressing these challenges, an interactive podcast program,

"Living with Type 1 Diabetes to Grown-Up"; is being developed with a one-year grant from the National Science and Technology Council. This continued project will span three years, employing a mixed-method research design for evaluation. Participants will be recruited from pediatric endocrinology and genetics clinics and wards across two medical centers in Northern Taiwan. In line with recommendations from prior reviewers, the study will incorporate a two-phased approach: the first phase is a quantitative study, structured around transitional theory and self-regulation theory using PRIDE steps. It adopts a double-blinded, randomized controlled experimental method with data collector and sham treatment participants blinded. Subjects will be randomly assigned to either the experimental group (N=44) or the active control group (N=44). Comparative analyses will focus on variations in disease control, emotional disturbance, confidence in self-management, self-care behaviors, diabetes knowledge, interpersonal disturbance, and family conflict at baseline, and post-interventions of immediate, 3-month, and 6-month periods. In the subsequent qualitative phase, 15-20 cases from the experimental group will be selected for in-depth interviews to evaluate the impact of the " Living with Type 1 Diabetes to GrownUp " interactive podcast program.

The outcomes of this research are anticipated to contribute significantly to the clinical management and technological intervention strategies for T1D adolescents in their transitional phase to adulthood.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of T1D by an endocrinologist before the age of 16 and a disease duration of >6months
* patients aged 16-25 years
* mean HbA1C level ≥7.5% one year before inclusion
* ability to communicate in Chinese or Mandarin
* patients who own smartphones with internet access
* patients who agreed to voice recording during a session explaining the treatment process
* patients who signed the informed consent form prior to participation; for minors, a legal representative must provide consent and sign the informed consent form.

Exclusion Criteria:

# T1D patients with other concomitant metabolic diseases, chromosomal aberrations, major illnesses, and cognitive impairment will be excluded from this study.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of HbA1C (%) in participants | Baseline and 3, 6months
  HbA1c from baseline, 3month and 6 months
percentage of self-monitored blood glucose readings within the 70-180 mg/dl range in Participants | Baseline and 3, 6months
  the percentage of self-monitored blood glucose levels within the optimal range of 70-180 mg/dL
Number of Hyperglycemic Events in Participants | Baseline and 3, 6months
  Number of events of each participant with blood sugar >200 mg/dl or" high" on glucometer, Ketoacidosis diagnosed
Number Hypoglycemic Events in Participants | Baseline and 3, 6months
  Number of events of each participant with blood sugar <60 mg/dl or "low" on glucometer, Hypoglycemia diagnosed

SECONDARY OUTCOMES:
Score of Diabetes Distress in Participants | Baseline and 3, 6months
  Change in Diabetes Distress Scale score over time.Diabetes Distress Scale (DDS): The original scale was developed by Polonsky et al. (2005). The Chinese version consists of 18 items across four subscales. Items are scored on a 4-point Likert scale ranging from 1 (no distress) to 4 (severely distressed), with higher scores indicating more severe emotional distress. Cronbach's α and test-retest reliability values of the DDS were 0.89 and 0.81, respectively (Liu et al., 2010).
Score of Diabetes Self-Managemen in Participants | Baseline and 3, 6months
  Perceived Diabetes Self-Management Scale (PDSMS):The original questionnaire was developed by Wallston et al. (2007). It consists of 8 items scored on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree),The translated questionnaire has content validity, Cronbach's α, and test-retest reliability values of 0.75, 0.93, and 0.97, respectively.
Score of Diabetes Self-care in Participants | Baseline and 3, 6months
  Self-care Behavior Assessment Scale: This scale was developed by Wang (2010) to measure self-care behaviors of adolescents with T1D. A total of 39 items are scored on a 5-point Likert scale ranging from 1 (not achieved at all) to 5 (completely achieved). The total score ranges from 39 to 195, with higher scores indicating better self-care behaviors. Cronbach's α and the content validity index (CVI) value based on content rating by experts are 0.87 and 0.92, respectively.
Score of Diabetes Knowledge in Participants | Baseline and 3, 6months
  Diabetes Knowledge Questionnaire (DKQ): The original questionnaire was developed by Garcia et al. (2001). The Chinese version comprises 24 items that are answered "Yes," "No" or "I don't know"; 1 point is awarded for each correct answer. The total score ranges from 0 to 24 points.reliability and Cronbach's α values of 0.78 and 0.89, respectively Hu et al.(2013)
Score of Interpersonal Distress in Participants | Baseline and 3, 6months
  Analyze the score changes in the "Diabetes-Related Interpersonal Distress" subscale within the Diabetes Distress Scale (as previously mentioned in the Diabetes Distress Scale score ).
Score of Diabetes-Related Family Conflict in Participants | Baseline and 3, 6months
  The Diabetes Family Conflict Scale-Revised (DFCS), revised by Hood et al. (2007), is used to assess family conflict and disagreements related to diabetes care in adolescents with T1D and their parents. The scale consists of 19 items and uses a 3-point scoring system: "Almost Never" scores 1 point, "Sometimes" scores 2 points, and "Almost Always" scores 3 points. Higher scores indicate more conflict. The DFCS has strong psychometric properties, with a Cronbach's α value of .95 for the adolescent version of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Tao Chiang, PhD, Study Director — Chang Gung University; Fu-Sung Lo, BSN, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang-Gung University and Chang-Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chiang YT, Lo FS, Yu HY, Chen CW, Moons P. Efficacy of the Online Interactive Podcast Program "Living With Type 1 Diabetes to Grown-Up": A Two-Arm Randomized Controlled Trial Protocol. J Diabetes Res. 2025 Sep 13;2025:4866975. doi: 10.1155/jdr/4866975. eCollection 2025. PMID 40978315